CLINICAL TRIAL: NCT02035553
Title: A Single Center, Double-Blind, Placebo-Controlled Study to Examine the Safety and Efficacy of Pimavanserin for the Treatment of Psychosis in Alzheimer's Disease
Brief Title: A Study of the Safety and Efficacy of Pimavanserin in Patients With Alzheimer's Disease Psychosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-019
Record Dates: First submitted 2014-01-13; First posted 2014-01-14 (Estimated); Results first posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-09

CONDITIONS: Alzheimer's Disease Psychosis
MeSH Terms: interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo, two tablets, once daily by mouth
  Interventions: Drug: Placebo
- Pimavanserin 40 mg (Experimental): Pimavanserin tartrate, 40 mg (two 20 mg tablets), once daily by mouth (equivalent to 34 mg free base pimavanserin)
  Interventions: Drug: Pimavanserin tartrate

INTERVENTIONS:
Drug: Pimavanserin tartrate — Pimavanserin tartrate, 40 mg (two 20 mg tablets), once daily by mouth (equivalent to 34 mg free base pimavanserin)
  Other Names: ACP-103
  Arms: Pimavanserin 40 mg
Drug: Placebo — Placebo, two tablets, once daily by mouth
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of pimavanserin 40 mg compared to placebo in patients with Alzheimer's disease psychosis.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 50 years of age or older with NINCDS-ADRDA defined possible or probable AD
* Patient must have psychotic symptoms that developed after the diagnosis of AD was established. These symptoms must include visual and/or auditory hallucinations, and/or delusions
* Patient must have been a nursing home resident for ≥ 4 weeks prior to randomization, not bedridden and expected to remain in the facility throughout the study
* Patient must have actively experienced and verbally communicated psychotic symptoms during the month prior to the Screening visit and weekly during the previous 2 weeks prior to Baseline
* If patient is on acetylcholinesterase inhibitor (AChEI) therapy and/or memantine, must be on stable doses for 3 months prior to the Baseline visit and during the study
* Patient is willing and able to provide informed consent. If the subject is unable to provide written consent due to the severity of dementia, consent must be given by a legally authorized representative

Exclusion Criteria:

* Patient has a history of significant psychotic disorders prior to or concomitantly with the diagnosis of Alzheimer's disease including, but not limited to, schizophrenia or bipolar disorder
* Patient is unable to communicate verbally
* Patient has current evidence of a serious and/or unstable cardiovascular, respiratory, gastrointestinal, renal, hematologic or other medical disorder, including cancer or malignancies, which would affect the patient's ability to participate in the study
* Patient has had a myocardial infarction in the last six months
* Patient has moderate to severe congestive heart failure
* Patient has any surgery planned during the screening, treatment, or follow-up periods that could interfere with participation in the study per the protocol assessments

Patients will be evaluated at screening to ensure that all criteria for study participation are met. These evaluations will include specific measures of psychosis severity, delirium, dementia, cardiovascular condition, and pregnancy status. Patients may be excluded from the study based on these assessments (and specifically if it is determined that their baseline health and psychiatric condition do not meet all protocol-specified entry criteria).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09-28 (Actual); Study Completion 2016-10-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- London, United Kingdom

REFERENCES:
- [Derived] Muhlbauer V, Mohler R, Dichter MN, Zuidema SU, Kopke S, Luijendijk HJ. Antipsychotics for agitation and psychosis in people with Alzheimer's disease and vascular dementia. Cochrane Database Syst Rev. 2021 Dec 17;12(12):CD013304. doi: 10.1002/14651858.CD013304.pub2. PMID 34918337
- [Derived] Ballard C, Banister C, Khan Z, Cummings J, Demos G, Coate B, Youakim JM, Owen R, Stankovic S; ADP Investigators. Evaluation of the safety, tolerability, and efficacy of pimavanserin versus placebo in patients with Alzheimer's disease psychosis: a phase 2, randomised, placebo-controlled, double-blind study. Lancet Neurol. 2018 Mar;17(3):213-222. doi: 10.1016/S1474-4422(18)30039-5. PMID 29452684

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Pimavanserin 40 mg
Started | 91 | 90
Completed | 73 | 67
Not Completed | 18 | 23
Not completed — Death (See All-Cause Mortality Table) | 0 | 1
Not completed — Adverse Event | 10 | 6
Not completed — Physician Decision | 3 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Non-compliance with Study Drug | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other Reason | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pimavanserin 40 mg | Total
Number analyzed (Participants) | 91 | 90 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 86.1 (5.96) | 85.7 (7.05) | 85.9 (6.51)
Age, Customized [Count of Participants; unit: Participants]
  Age: <=85 | 41 | 41 | 82
  Age: >85 | 50 | 49 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 73 | 146
  Male | 18 | 17 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 91 | 90 | 181
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 0 | 3 | 3
  Race: Black or African American | 1 | 3 | 4
  Race: White | 89 | 84 | 173
  Race: Other | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 91 | 90 | 181

OUTCOME MEASURES:

1. Primary Outcome: Antipsychotic Efficacy
Description: Change from Baseline to Day 43 in the Neuropsychiatric Inventory-Nursing Home Version (NPI-NH) psychosis score (Delusions [Domain A]+Hallucinations [Domain B]) in the Full Analysis Set (FAS). The NPI-NH is a questionnaire that quantifies behavioral changes in dementia in nursing home patients and evaluates 12 behavioral domains. For each of the 12 behavioral domains the Frequency (scale:1=occasionally to 4=very frequently) is multiplied by the Severity (scale:1=Mild to 3=Severe) to obtain a domain score (frequency x severity), The NPI-NH Psychosis Subscale consists of the two domains of Delusions and Hallucinations, calculated by adding the Individual domain scores, to yield a possible total score of 0 to 24. Lower scores correspond to less severity. A negative change score from baseline indicates improvement.
Time Frame: Day 43
Population: All randomized subjects who received at least one dose of study treatment and have both a Baseline and at least one post-Baseline NPI-NH psychosis score evaluation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on the NPI-NH scale
Arm/Group | Placebo | Pimavanserin 40 mg
Number analyzed (Participants) | 91 | 87
Score on the NPI-NH scale | -1.93 [-3.18 to -0.67] | -3.76 [-5.05 to -2.47]
Statistical Analysis 1: Comparison: Placebo vs Pimavanserin 40 mg; Test type: Superiority; p = 0.0451, Mixed Models Analysis; Diff in MMRM LSM = -1.84, 95% CI 2-sided [-3.64 to -0.04]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: From the time the informed consent was signed, adverse events were recorded in the subject's source documents and entered into the appropriate eCRF pages at the Screening visit, at visits on Study Days 1, 15, 29, 43, 64 and Day 85, and at the 4-week follow-up phone call.
Arm/Group | Placebo | Pimavanserin 40 mg
All-Cause Mortality (participants affected / at risk) | 4/91 | 4/90
Serious Adverse Events (participants affected / at risk) | 10/91 | 15/90
Other Adverse Events (participants affected / at risk) | 70/91 | 67/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=91) | Pimavanserin 40 mg (N=90)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) — General disorders and administration site conditions
Pneumonia (Infections and infestations) | 2 (2) | 2 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Malignant neoplasm of thorax (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Aggression (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=91) | Pimavanserin 40 mg (N=90)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 9 (9)
Oedema peripheral (General disorders) | 2 (2) | 7 (7) — General disorders and administration site conditions
Urinary tract infection (Infections and infestations) | 25 (36) | 18 (27)
Lower respiratory tract infection (Infections and infestations) | 12 (13) | 13 (15)
Cellulitis (Infections and infestations) | 3 (3) | 6 (7)
Fall (Injury, poisoning and procedural complications) | 21 (35) | 20 (39)
Contusion (Injury, poisoning and procedural complications) | 14 (17) | 11 (16)
Laceration (Injury, poisoning and procedural complications) | 5 (6) | 3 (3)
Blood urea increased (Investigations) | 8 (8) | 7 (7)
Blood potassium increased (Investigations) | 3 (3) | 5 (5)
Blood lactate dehydrogenase increase (Investigations) | 10 (10) | 4 (4)
Blood alkaline phosphatase increased (Investigations) | 8 (8) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (11) | 4 (4)
Somnolence (Nervous system disorders) | 7 (7) | 3 (3)
Agitation (Psychiatric disorders) | 13 (13) | 19 (19)
Aggression (Psychiatric disorders) | 4 (4) | 9 (10)
Anxiety (Psychiatric disorders) | 2 (2) | 5 (5)
Behavioural and psychiatric symptoms of dementia (Psychiatric disorders) | 2 (2) | 5 (6)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to his/her own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the sponsor for review and comment. The sponsor has 60 days to review and comment.